CLINICAL TRIAL: NCT05646017
Title: Effect of the Greatest Spanish Heatwave Over Glycemic Control in Adult Patients With Type 1 Diabetes
Brief Title: Effect of Heatwave Over Glycemic Control in Patients With T1D
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: C-566
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes patients: Type 1 diabetes patients using intermittently continuous glucose monitoring during the Spanish greatest heatwave in Castilla-La Mancha (Spain).
  Interventions: Device: Intermittenly scanned continuous glucose monitoring

INTERVENTIONS:
Device: Intermittenly scanned continuous glucose monitoring — Use of Intermittenly scanned continuous glucose monitoring (FreeStyle Libre)
  Other Names: FreeStyle Libre; isCGM; FSL

SUMMARY:
Observational study about effect of the greatest Spanish heatwave over glycemic contro in adult patients with type 1 Diabetes mellitus.

DETAILED DESCRIPTION:
Cross-sectional retrospective analysis of all patients with T1D in Castilla-La Mancha (south-central Spanish region) using intermittently scanned continuous glucose monitoring (isCGM). Glycometric data obtained through deidentified downloads from isCGM´s webpage. Primary outcome was time in range (TIR) 3.0-10 mmol/L (70-180 mg/d) change after the heatwave. Data analysis is conducted using SPSS (Chicago, IL) statistics software. Results are presented as mean ± SD values or percentages. A paired Student's t-test or a Wilcoxon signed-rank test were used for the analysis of differences. Comparisons between proportions were analyzed using a chi-squared test. A P value < 0.05 was considered statistically significant. The protocol was approved by the reference Castilla-La Mancha Public Health Institute Ethic Committee.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Older than 18 years old
* Using intermittently scanned continuous glucose monitoring (isCGM)
* Paired active isCGM data from the heatwave period and two consecutive weeks

Exclusion Criteria:

* Younger than 18 years old
* Not using intermittently scanned continuous glucose monitoring
* Not having active paired isCGM data from the analyzed periods

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult type 1 diabetes patients using intermittently scanned continuous glucose monitoring during and after the greatest Spanish heatwave.
Sampling Method: Non-Probability Sample
Enrollment: 2701 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Time in range | 14 days
  Change in Time in range (TIR) 3.0-10 mmol/L (70-180 mg/d) of interstitial glucose from the heatwave period to 14 days after its end

SECONDARY OUTCOMES:
Change in Adherence to Flash 1 | 14 days
  Change in Time of use of intermittently scanned continuous glucose monitoring (% possible time of use) from the heatwave period to 14 days after its end
Change in Adherence to Flash 2 | 14 days
  Change in Number of intermittently scanned continuous glucose monitoring daily scanning (number of scans/day) from the heatwave period to 14 days after its end
Change in Time below range 1 (TBR1) | 14 days
  Change in Time bellow range <3.9 mmol/L (<70 mg/dL) of the interstitial glucose from the heatwave period to 14 days after its endfrom the heatwave period to 14 days after its end
Change in Time below range 2 (TBR2) | 14 days
  Change in Time bellow range <3 mmol/L (<54 mg/dL) of the interstitial glucose from the heatwave period to 14 days after its end
Change in Time above range 1 (TAR1) | 14 days
  Change in Time above range >10 mmol/L(>180 mg/dL) of the interstitial glucose from the heatwave period to 14 days after its end
Change in Time above range 2 (TAR2) | 14 days
  Change in Time above range >13.9 mmol/L (>250 mg/dL) of the interstitial glucose from the heatwave period to 14 days after its end
Change in Coefficient of variation percentage (CV) | 14 days
  Change in Coefficient of variation percentage of interstitial glucose from the heatwave period to 14 days after its end
Change in Glucose management index | 14 days
  Change in Glucose management index of interstitial glucose from the heatwave period to 14 days after its end
Change in Time in hypoglycemia | 14 days
  Change in Daily time in hypoglycemia (<3.9 mmol/L, <70 mg/dL) of interstitical glucose from the heatwave period to 14 days after its end
Change in Hypoglycemia frequency | 14 days
  Change in Number of daily hypoglycemic events (<3.9 mmol/L, <70 mg/dL) of interstitical glucose from the heatwave period to 14 days after its end

OTHER OUTCOMES:
Change in Percentage of patients attaining the the International Consensus on Time in Range (ICTR) goals | 14 days
  Change in Percentage of patients (from total) attaining TIR>70%, TBR1<4%, TBR2<1%, TAR1<25%, TAR2<5% and CV <36% from the heatwave period to 14 days after its end

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - La Mancha-Centro Hospital, Alcázar de San Juan, Ciudad Real
  - Santa Barbara Hospital, Puertollano, Ciudad Real
  - Valdepeñas General Hospital, Valdepeñas, Ciudad Real
  - Virgen del Prado Hospital, Talavera de la Reina, Toledo
  - Albacete University Hospital, Albacete
  - Ciudad Real General University Hospital, Ciudad Real
  - Virgen de la Luz University Hospital, Cuenca
  - Guadalajara University Hospital, Guadalajara
  - Toledo University Hospital, Toledo

IPD SHARING:
Plan to Share IPD: No
Under other researchers request.

REFERENCES:
- [Background] Song X, Jiang L, Zhang D, Wang X, Ma Y, Hu Y, Tang J, Li X, Huang W, Meng Y, Shi A, Feng Y, Zhang Y. Impact of short-term exposure to extreme temperatures on diabetes mellitus morbidity and mortality? A systematic review and meta-analysis. Environ Sci Pollut Res Int. 2021 Nov;28(41):58035-58049. doi: 10.1007/s11356-021-14568-0. Epub 2021 Jun 8. PMID 34105073
- [Background] Moon J. The effect of the heatwave on the morbidity and mortality of diabetes patients; a meta-analysis for the era of the climate crisis. Environ Res. 2021 Apr;195:110762. doi: 10.1016/j.envres.2021.110762. Epub 2021 Jan 27. PMID 33515577
- [Background] Xu Z, Tong S, Cheng J, Crooks JL, Xiang H, Li X, Huang C, Hu W. Heatwaves and diabetes in Brisbane, Australia: a population-based retrospective cohort study. Int J Epidemiol. 2019 Aug 1;48(4):1091-1100. doi: 10.1093/ije/dyz048. PMID 30927429
- [Result] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- See also: Spanish National Weather Agency — https://www.aemet.es/es/serviciosclimaticos/cambio_climat